CLINICAL TRIAL: NCT01423331
Title: An Evaluation and Factor Analysis for Maternal Mental Health - The Analytic Study of the Shin Kong Wu Ho-Su Memorial Hospital
Brief Title: An Evaluation and Factor Analysis for Maternal Mental Health
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Principal Investigator, Yieh-Loong Tsai, Gynecologist, Shin Kong Wu Ho-Su Memorial Hospital
Other Study IDs: 20110409R
Record Dates: First submitted 2011-08-24; First posted 2011-08-25 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Postpartum Depression
Keywords: Postpartum depression; maternal mental health
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An Evaluation and Factor Analysis for Maternal Mental Health - The Analytic Study of the Shin Kong Wu Ho-Su Memorial Hospital

- Objectives：

1. To construct a screening tool for domestic maternal mental health
2. To expect to find the screening timing for early assessment or intervention of domestic maternal mental health status.
3. To explore the impact of domestic maternal mental health factors.

DETAILED DESCRIPTION:
-Study Design： This project will be conducted at the Shin Kong Memorial Hospital for pregnant women or mothers within six months after birth, with the base of existing domestic and foreign screening tools for postpartum depression and the related scale modeled, and select respective women during different pregnant period and after birth as postpartum study, by longitudinal study and cross-sectional study of the advantages to be able to plan time for up to twelve months of data collection, able to undertake within-subjects comparison and the between-subjects comparison, to view depression during pregnancy , pregnancy depression, postpartum blues, postpartum depression, postpartum psychosis such as prevalence, risk factors or any other factors.

To establish the screening tool and screening time for national early assessment of maternal mental health status of women in pregnancy and after birth.

-Effect：

1. Expected to construct the applicable domestic early assessment screening or intervention time of maternal mental health status.
2. Expected to develop different screening tools for a domestic early assessment of the maternal mental health status.
3. Expected to identify the important factors of maternal depression to provide a reference for locking in a high risk group for early intervention.
4. The implementation of women's health policy on mental health care of pregnant women with specific feasible approach.
5. To provide mental health counseling, the implementation of the operation of the network of community resources to reduce maternal stress in coping to new life.

ELIGIBILITY:
Inclusion Criteria:

* the pregnant women or mothers within six months after birth

Exclusion Criteria:

* Minor

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the pregnant women or mothers within six months after birth
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yieh-Loong Tsai, Study Chair — Shin Kong Wu Ho-Su Memorial Hospital